CLINICAL TRIAL: NCT05788770
Title: Preoperative CT-imaging with Patient-specific Computer Simulation in Transcatheter Aortic Valve Replacement: a Randomized Controlled Trial
Brief Title: Preoperative CT-imaging with Patient-specific Computer Simulation in Transcatheter Aortic Valve Replacement
Acronym: GUIDE-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Romy Hegeman (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Romy Hegeman, Research Coordinator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL77697.100.21
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Multicenter, multinational, randomized controlled, open-label, trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FEops HEARTGuide (Experimental): Device selection using FEops HEARTGuide: 3D anatomical analysis and simulation of transcatheter aortic valve prosthesis prior to procedure based on computed tomography.
  Interventions: Other: FEops HEARTGuide
- Standard transcatheter aortic valve implantation (no FEops HEARTGuide) (No Intervention): Control: standard of care, CT based device selection.

INTERVENTIONS:
Other: FEops HEARTGuide — FEops HEARTGuide added to routine preoperative CT imaging. Results of the computer modelling will be discussed with TAVR implanting team prior to and during the procedure.
  Arms: FEops HEARTGuide

SUMMARY:
Combining routine preoperative CT imaging with patient-specific computer modelling predicts the interaction between different sizes of transcatheter aortic valve replacement devices at different implantation depths and the patient's unique anatomy (including post-implantation deformation) allowing preoperative evaluation of the risk for paravalvular leakage and conduction disorders.

The objective of this randomized controlled trial is to evaluate whether pre-operative CT-imaging with advanced computer modelling and simulation (FEops HEARTguide™) adequately predicts procedural outcomes in TAVR procedures, whether it leads to changes of preoperative decisions and whether or not this leads to improved outcome in TAVR procedures.

ELIGIBILITY:
Inclusion Criteria:

* Primary symptomatic severe aortic valve stenosis
* Accepted for TAVR, either by transfemoral, transsubclavian or transapical access
* Plan to implant one of the following transcatheter heart valves for which FEops HEARTguide™ is available (CoreValve™ Evolut™ R, and Evolut™ PRO and Evolut™ PRO+ (Medtronic, Minnesota, USA), ACURATE neo™ and ACURATE neo 2™ (Boston Scientific, Marlborough, MA, USA)
* Informed consent

Exclusion Criteria:a potential subject who meets any of the following criteria will be excluded from participation in this study before randomization:

* Previous surgical aortic valve replacement
* Permanent pacemaker at baseline
* Emergency procedure
* Poor CT image quality (disabling computer-simulation, i.e. generation of 3D anatomical models will not be possible with poor CT image quality), for example because of motion artifacts due to the presence of other implanted devices affecting the region of interest
* Patient who did not agree to the informed consent and/or refused to participate
* Patient unable to understand the informed consent/study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mild to severe paravalvular regurgitation | 30-days

SECONDARY OUTCOMES:
Incidence of new conduction disorder (new-onset left bundle branch block or new-onset atrioventricular block) | 30 days after TAVI
Need for permanent pacemaker implantation | 30 days after TAVI
Preoperative valve size selection | Preprocedural
Final valve size | Perprocedural
Target implantation depth | Preprocedural
Final implantation depth | Perprocedural
Change of preoperative decision in choice of default transcather heart valve | Preprocedural
Change of preoperative decision in valve size selection | Preprocedural
Change of preoperative decision in target implantation depth | Preprocedural
Failure to implant valve | Preprocedural
Composite endpoint of major adverse cardiac and cerebrovascular events (MACCE) | 30 days after TAVI
  Including mortality, stroke, life-threatening bleeding, major vascular complications, valve-related dysfunction requiring repeat procedure (TAVR or SAVR), according to the VARC-3 criteria
Quality of life assessed by the EuroQol questionnaire | 90 days after TAVI
  EuroQol-5 Dimensions-5 Levels, lower levels refer to better outcomes. Visual analog scale (0-100). Higher scores refer to a better outcome.
Quality of life assessed by the Kansas City Cardiomyopathy Questionnaire | 90 days after TAVI
  All scores are represented on a 0-to-100-point scale. Higher score refers to preferabel outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Klein, MD, PhD, Principal Investigator — St. Antonius Hospital; Martin Swaans, MD, PhD, Principal Investigator — St. Antonius Hospital; Prof. Jurriën ten Berg, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (2):
- Vienna General Hospital, Vienna, Austria
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided